CLINICAL TRIAL: NCT05276739
Title: Determining the Role of Photic and Non-photic Time Cues in Resetting Circadian Rhythms in Humans
Brief Title: Role of Photic and Non-photic Time Cues in Resetting Circadian Rhythms
Acronym: LipidPRC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shadab A Rahman, Assistant Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2021P000757
Record Dates: First submitted 2022-03-03; First posted 2022-03-11 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Light Exposure; Meal Timing

STUDY DESIGN:
Intervention Model Description: 3 condition, parallel arm randomized control trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bright light (Experimental): Participants will receive a 6.5-hour 10,000 lux light pulse (4100K fluorescent light) centered within the 16-hour wake episode (start 4.75 hour after wake and end 11.25 hour after wake). Participants will receive 4 identical meals (equal calories and macronutrient content), over a 12-hour interval (meals at 2, 6, 10, and 14 hours after waking) centered within the 16-hour wake episode.
  Interventions: Behavioral: Bright Light; Behavioral: 12-h meal window
- Time-restricted eating (Experimental): Participants will consume 4 identical meals, as in the other groups, except that the meal window will be restricted to 6.5 hours instead of 12 hours (meals at 4.75, 6.9, 9.1, 11.25 hours after waking) centered within the 16-hour wake episode. Participants will remain in dim light (<3 lux) throughout the 16-hour wake episode.
  Interventions: Behavioral: Time-restricted eating; Behavioral: Dim light
- Control (Sham Comparator): Participants will receive 4 identical meals (equal calories and macronutrient content), over a 12-hour interval (meals at 2, 6, 10, and 14 hours after waking) centered within the 16-hour wake episode. Participants will remain in dim light (<3 lux) throughout the 16-hour wake episode.
  Interventions: Behavioral: Dim light; Behavioral: 12-h meal window

INTERVENTIONS:
Behavioral: Bright Light — 6.5-hour 10,000 lux light pulse (4100K fluorescent light) centered within the 16-hour wake episode (start 4.75 hour after wake and end 11.25 hour after wake).
  Arms: Bright light
Behavioral: Time-restricted eating — 6.5-hour restricted meal window (4 meals at 4.75, 6.9, 9.1, 11.25 hours after waking) centered within the 16-hour wake episode.
  Arms: Time-restricted eating
Behavioral: Dim light — dim light (<3 lux) throughout the 16-hour wake episode
  Arms: Control; Time-restricted eating
Behavioral: 12-h meal window — 12-hour restricted meal window (4 meals at 2, 6, 10, and 14 hours after waking) centered within the 16-hour wake episode.
  Arms: Bright light; Control

SUMMARY:
The aim of this study is to determine the principal time cue (light or meals) for resetting circadian rhythms in melatonin and metabolic outcomes.

DETAILED DESCRIPTION:
The objective of this proposal is to construct and compare PRCs describing the relationship between the timing of light exposure and meals across the 24-hour day and the size and direction of shift in circadian rhythms of circulating lipids and melatonin in humans. Completion of the work will provide mechanistic insight on the role of photic and non-photic cues mediating entrainment of circadian rhythms in humans besides that of melatonin. In this proposal, we will use the same experimental paradigm that we have successfully used previously to characterize and compare PRCs for shifts in melatonin in response to light exposure of different durations and spectra, and as used in our pilot trials demonstrating a robust PRC of lipid circadian rhythms in response to combined photic and non-photic stimuli across the day. We will achieve our objective using a randomized controlled trial in young healthy adults (n=48, 18-30 years) that systematically manipulates the timing of 6.5-hour bright light exposure and 6.5-hour time restricted eating across the 24-hour circadian cycle to specifically:

Aim 1: Determine if light is the primary time cue for resetting melatonin but not lipid circadian rhythms. Hypothesis: The resetting response of circadian rhythms in melatonin but not cholesterol and triglycerides is dependent upon the circadian phase at which a 6.5-hour bright light exposure occurs.

Aim 2: Determine if meal timing is the primary time cue for resetting lipid but not melatonin circadian rhythms. Hypothesis: The resetting response of circadian rhythms in cholesterol and triglycerides but not melatonin is dependent upon the circadian phase at which a 6.5-hour time restricted eating occurs.

Aim 3 (Exploratory): Evaluate the acute effects of eating across the 24-hour day on circulating lipid levels. Hypothesis: The acute effects of 6.5-hour time restricted eating on circulating cholesterol and triglycerides levels are dependent on the circadian phase at which meals are eaten.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-30 years
* Healthy (no medical, psychiatric or sleep disorders;
* Non-smoking for at least 6 months;
* Body Mass Index of >18 or <30 kg/m2;
* Able to maintain 8-hour consistent sleep schedule during the study
* Able to refrain from caffeine, alcohol, medication and supplements during the study

Exclusion Criteria:

* History of alcohol or substance abuse;
* Positive result on drugs of abuse urine toxicology;
* Current or past history of sleep disorders, including but not limited to obstructive sleep apnea, narcolepsy, insomnia, or any significant sleep complaint
* Psychiatric disorder, or first degree relative with a psychiatric disorder
* Recent acute or chronic medical disorder
* Use of drugs or medication (birth control OK) likely to affect sleep, alertness or light sensitivity, as determined by the investigators
* Visual disorder, including but not limited to color blindness, or family history of glaucoma
* Pregnancy or lactation
* Shift work (past 3 years)
* Transmeridian travel (2 or more time zones) in the past 3 months
* Any other reason as determine by the Principal Investigator

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-07-29 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Amplitude of Phase Response Curve of melatonin | 24 hours
  Amplitude of phase response curve of melatonin derived by fitting a sinusoidal regression to the individual phase shift data across ~24 hours
Amplitude of Phase Response Curve of triglyceride | 24 hours
  Amplitude of phase response curve of triglyceride derived by fitting a sinusoidal regression to the individual phase shift data across ~24 hours
Amplitude of Phase Response Curve of cholesterol | 24 hours
  Amplitude of phase response curve of cholesterol derived by fitting a sinusoidal regression to the individual phase shift data across ~24 hours

SECONDARY OUTCOMES:
Area under the curve (AUC) of melatonin | 6.5 hours during intervention
  AUC of melatonin
Area under the curve (AUC) of triglyceride | 6.5 hours during intervention
  AUC of triglyceride
Area under the curve (AUC) of cholesterol | 6.5 hours during intervention
  AUC of cholesterol

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No